CLINICAL TRIAL: NCT01212991
Title: PREVAIL: A MULTINATIONAL PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED EFFICACY AND SAFETY STUDY OF ORAL MDV3100 IN CHEMOTHERAPY-NAÏVE PATIENTS WITH PROGRESSIVE METASTATIC PROSTATE CANCER WHO HAVE FAILED ANDROGEN DEPRIVATION THERAPY
Brief Title: A Safety and Efficacy Study of Oral MDV3100 in Chemotherapy-Naive Patients With Progressive Metastatic Prostate Cancer
Acronym: PREVAIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDV3100-03; 2010-020821-41 (EudraCT Number); C3431003 (Other: Alias Study Number)
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: Progressive Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzalutamide (Experimental)
  Interventions: Drug: Enzalutamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enzalutamide — Participants received enzalutamide 160 mg, administered as four 40-mg capsules, once per day by mouth. Study drug treatment continued until disease progression (evidence of radiographic progression, a skeletal-related event, or clinical progression) and the initiation of a cytotoxic chemotherapy or an investigational agent, unacceptable toxicity, or withdrawal.
  Arms: Enzalutamide
Drug: Placebo — Participants received placebo, administered as four capsules, once per day by mouth. Study drug treatment continued until disease progression (evidence of radiographic progression, a skeletal-related event, or clinical progression) and the initiation of a cytotoxic chemotherapy or an investigational agent, unacceptable toxicity, or withdrawal.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the benefit of enzalutamide versus placebo as assessed by overall survival and progression-free survival in patients with progressive metastatic prostate cancer who have failed androgen deprivation therapy but not yet received chemotherapy.

ELIGIBILITY:
Randomized, Double Blind Treatment Period:

Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Ongoing androgen deprivation therapy with a GnRH analogue or bilateral orchiectomy
* Progressive disease despite androgen deprivation therapy as defined by rising PSA levels or progressive soft tissue or bony disease
* No prior treatment with cytotoxic chemotherapy
* Asymptomatic or mildly symptomatic from prostate cancer

Exclusion Criteria:

* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment
* Known or suspected brain metastasis or active leptomeningeal disease
* History of another malignancy within the previous 5 years other than curatively treated non-melanomatous skin cancer

Open-Label Treatment Period:

The following inclusion criteria apply to patients receiving enzalutamide or placebo during double-blind treatment.

Eligible patients must meet all inclusion criteria.

* Received randomized double-blind treatment in PREVAIL;
* Open-label day 1 visit is within 6 months after this amendment is approved and becomes effective at the study site;
* Is willing to maintain androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) agonist/antagonist or has had a bilateral orchiectomy;

The exclusion criteria apply only to patients starting new treatment with enzalutamide after receiving placebo as randomized treatment. Each patient must not meet any of the following criteria:

* Has taken commercially available enzalutamide (Xtandi);
* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment
* Known or suspected brain metastasis or active leptomeningeal disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1717 (Actual)
Dates: Start 2010-09-16 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (267):
- United States (64):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Cancer Certer-North Campus, Tucson, Arizona
  - Cancer Center Oncology Medical Group, La Mesa, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC&USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center / Investigational Drug Services, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center Drug Information Center Department of Pharmaceutical Services, Los Angeles, California
  - UCLA Clark Urology Clinic, Los Angeles, California
  - North County Oncology Medical Clinic, Inc, Oceanside, California
  - UC Davis Medical Center, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Medical Oncology Associates-SD, San Diego, California
  - Sharp Memorial Hospital Investigational Pharmacy, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Anschutz Cancer Center Pavilion Pharmacy, Aurora, Colorado
  - University of Colorado Hospital, Anschutz Cancer Pavilion, Aurora, Colorado
  - Lynn Cancer Institute Center for Hematology Oncology, Boca Raton, Florida
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Jewish Hospital & St. Mary's Healthcare, Inc., Louisville, Kentucky
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaoness Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish St. Peters Hospital, City of Saint Peters, Missouri
  - Barnes-Jewish West County Hospital, Creve Coeur, Missouri
  - BJH Pharmacy, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - The Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cancer Centers of North Carolina, Cary, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Levine Cancer Institute - Main, Charlotte, North Carolina
  - Levine Cancer Institute - Southpark, Charlotte, North Carolina
  - Levine Cancer Institute - University, Charlotte, North Carolina
  - Levine Cancer Institute - Ballantyne, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Investigational Chemotherapy Services, Durham, North Carolina
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Portland VA Medical Center Laboratory, Portland, Oregon
  - Abramson Cancer Center of the University of Pennsylvania at Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Hematology / Oncology MUSC Hollings Cancer Center, Charleston, South Carolina
  - Medical University of South Carolina - Urology Services, Charleston, South Carolina
  - MUSC Department of Radiology, Charleston, South Carolina
  - MUSC Urology Ambulatory Care, Charleston, South Carolina
  - MUSC Hematology / Oncology Medical Specialty Associates, East Cooper Medical Arts Center 3rd Floor, Mt. Pleasant, South Carolina
  - MUSC Urology Medical Specialty Associates, East Cooper Medical Arts Center 3rd Floor, Mt. Pleasant, South Carolina
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (42):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Private Hospital, Kogarah, New South Wales
  - Lismore Base Hospital, Lismore Cancer Care and Haematology Unit, Lismore, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - North Coast Cancer Institute, Port Macquarie, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Department of Medical Oncology, St Leonards, New South Wales
  - Sydney Adventist Hospital, Sydney, New South Wales
  - Australian Clinical Trials Pty Ltd, Wahroonga, New South Wales
  - SAN Pathology, Wahroonga, New South Wales
  - SAN Radiology, Wahroonga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Heart Care Partners, Auchenflower, Queensland
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - River City Pharmacy, Auchenflower, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - University of Queensland Centre for Clinical Research (UQCCR), Herston, Queensland
  - Nuclear Medicine and Imaging Department, Herston, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Mater Private Cardiology, South Brisbane, Queensland
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - APHS Pharmacy, Kurralta Park, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Cancer Care SA Pty Ltd, Kurralta Park, South Australia
  - Bendigo Health, Bendigo Hospital, Bendigo, Victoria
  - Bendigo Health Medical Imaging, Bendigo, Victoria
  - Eastern Health, Box Hill, Victoria
  - MIA Box Hill Radiology, Box Hill, Victoria
  - Oncology Eastern Clinical Research Unit (ECRU), Box Hill, Victoria
  - Pharmacy Department, Box Hill, Victoria
  - Cabrini Hospital Brighton, Brighton, Victoria
  - Monash Health Translation Precinct, Clayton, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Barwon Health, Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Cabrini Radiology, Malvern, Victoria
  - MDI Chemer, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Austria (4):
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Ordination Dr. Fink, Salzburg
  - Salzburger Universitatsklinikum, Salzburg
  - Medizinische Universitaet Wien, Vienna
- Belgium (6):
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Sint-Lucas, Ghent
  - Jessaziekenhuis, Hasselt
  - AZ Groeninge, Campus KL, Kortrijk
  - UZ Leuven - University Hospital Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege-Urologie, Liège
- Canada (19):
  - Alberta Health Services - Cancer Care, Tom Baker Cancer Centre, Calgary, Alberta
  - Tom Baker Cancer Centre - Holy Cross Site, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Sindi Ahluwalia Hawkins, Centre for the Southern Interior, Kelowna, British Columbia
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - Vancouver Island Health Authority-Royal Jubilee Hospital Medical Imaging, Victoria, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - Manitoba Prostate Centre, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Nova Scotia Cancer Centre., Halifax, Nova Scotia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London RegCancer Program, London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, General Campus, Ottawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - CHU de Quebec - L'Hotel-Dieu de Quebec, Québec, Quebec
  - Centre de recherche clinique el evaluative en oncologie (CRCEO), Québec, Quebec
- Denmark (6):
  - Aalborg Hospital Nord, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Frederiksberg Hospital, Frederiksberg
  - Herlev Hospital, Herlev
  - Roskilde Sygehus, Roskilde
- Finland (4):
  - Docrates Clinic, Helsinki
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- France (17):
  - Hopital Civil, Strasbourg, Alsace
  - Centre Eugene Marquis-Service d'Oncologie Medicale, Rennes, Brittany Region
  - Institut Bergonie, Bordeaux, Nouvelle-Aquitaine
  - ICO Paul Papin, Angers
  - Clinique Rhone Durance, Avignon
  - Institut Bergonie, Bordeaux
  - CHD Vendee, La Roche-sur-Yon
  - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Groupe Hospitalier La Pitie Salpetriere, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Centre de Recherche Clinique, Saint-Herblain
  - HIA Begin, Service de Medecine Interne et Oncologie, Saint-Mandé
  - Institut de Cancerologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Clinique Pasteur, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (13):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Charite-Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Staedtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitaetsklinikum Carl Gustav Carus Dresden an der, Dresden
  - Martini-Klinik am UKE Gmbh, Hamburg
  - Urologikum Hamburg, Hamburg
  - Universitaetsklinikum Heidelberg, Klinik Fuer Urologie, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg/Saar
  - Universitaetsklinikum Mannheim, Klinik fuer Urologie, Mannheim
  - Universitaetsklinikum Muenster, Münster
  - Universitaetsklinikum Tuebingen, Universitaetsklinik fuer Urologie, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - Kliniken Nordoberpfalz AG, Klinikum Weiden, Weiden in Der Oberpfalz
- Israel (5):
  - Assaf Harofe Medical Center, Beer Yaakov
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
- Italy (6):
  - Azienda Socio Sanitaria Territoriale di Cremona, Cremona, CR
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola, FC
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, TO
  - Azienda USL8-Presidio Ospedaliero S.Donato, Arezzo
  - Ospedale G.B. Morgagni, Forlì
  - Azienda Ospedaliera San. Camillo Forlanini, Rome
- Japan (21):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Tokushima University Hospital, Tokushima, Tokushima
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Cancer Institute Hospital, Koutou-ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Keio University Hospital, Shinjyuku-ku, Tokyo
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
  - Chiba Cancer Center, Chiba
  - Kyoto University Hospital, Kyoto
  - Niigata University Medical and Dental Hospital, Niigata
  - Osaka City University Hospital, Osaka
  - Jikei University Hospital, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata
- Lithuania (2):
  - Klaipeda University Hospital, Klaipėda
  - Division of Oncourology, National Cancer Institute, Vilnius
- Netherlands (4):
  - Vrije Universiteit Medical Center, Department of Medical Oncology, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - University Medical Center Groningen, Department of Urology, Groningen
  - UMC St. Radboud, Nijmegen
- Poland (6):
  - Wielkopolskie Centrum Onkologii, Poznan, Greater Poland Voivodeship
  - EMC Instytut Medyczny S.A., Wroclaw, Lower Silesian Voivodeship
  - Apteka Szpitalna, Gdansk, Pomeranian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej, Mysłowice, Silesian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Tramatologii im. M.Kopernika w Lodzi, Lodz, Łódź Voivodeship
- Russia (4):
  - Russian Academy of Medical Sciences Institution, Moscow
  - North-Western State Medical University named after I.I.Mechnikov of the Ministry of Healthcare, Saint Petersburg
  - State Educational Institution of Higher Professional Education, Saint Petersburg
  - State healthcare institute, Saint Petersburg
- Singapore (2):
  - Department of Urology, National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Slovakia (6):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta B. bystrica, Banská Bystrica
  - CUIMED s.r.o., Bratislava
  - Univerzitna Nemocnica Martin, Martin
  - UROEXAM, spol. s r.o. urologicka ambulancia, Nitra
  - Poliklinika Sekcov, wesper, s.r.o., Prešov
  - UROCENTRUM MILAB s.r.o., Prešov
- South Korea (7):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-eup, Hwasun-gun, Jeollanam-do
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Asan Medical Center, Songpa-gu, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
- Spain (11):
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario German Trias i Pujol, Badalona, Barcelona
  - Althaia Xarxa Asistencial Manresa, Manresa, Barcelona
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Corporacio Sanitaria Parc Tauli, Sabadell(Barcelona)
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Malmo
  - Orebro University Hospital, Örebro
  - Karolinska University Hospital Solna, Stockholm
  - Umea University Hospital, Umeå
- United Kingdom (13):
  - Bishops Wood Hospital, Northwood, Middlesex
  - Mount Vernon Hospital, Northwood, Middlesex
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - Royal Marsden Hospital, Sutton, Surrey
  - Northern Centre for Cancer Care, Newcastle upon Tyne, TYNE and WEAR
  - Velindre Cancer Centre, Cardiff, Wales
  - Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral, Merseyside
  - Clinical Investigations and Research Unit, Royal Sussex County Hospital, Brighton, East Sussex
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Edinburgh Cancer Centre, Edinburgh
  - University College London Hospital NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Cella D, Ganguli A, Turnbull J, Rohay J, Morlock R. US Population Reference Values for Health-Related Quality of Life Questionnaires Based on Demographics of Patients with Prostate Cancer. Adv Ther. 2022 Aug;39(8):3696-3710. doi: 10.1007/s12325-022-02204-3. Epub 2022 Jun 22. PMID 35731340
- [Derived] Joshua AM, Armstrong A, Crumbaker M, Scher HI, de Bono J, Tombal B, Hussain M, Sternberg CN, Gillessen S, Carles J, Fizazi K, Lin P, Duggan W, Sugg J, Russell D, Beer TM. Statin and metformin use and outcomes in patients with castration-resistant prostate cancer treated with enzalutamide: A meta-analysis of AFFIRM, PREVAIL and PROSPER. Eur J Cancer. 2022 Jul;170:285-295. doi: 10.1016/j.ejca.2022.04.005. Epub 2022 May 26. PMID 35643841
- [Derived] Tombal BF, Freedland SJ, Armstrong AJ, Beer TM, Stenzl A, Sternberg CN, Hussain M, Ganguli A, Ramaswamy K, Bhadauria H, Ivanescu C, Turnbull J, Holmstrom S, Saad F. Impact of enzalutamide on patient-reported fatigue in patients with prostate cancer: data from the pivotal clinical trials. Prostate Cancer Prostatic Dis. 2022 Feb;25(2):288-295. doi: 10.1038/s41391-021-00447-9. Epub 2021 Sep 13. PMID 34518652
- [Derived] Armstrong AJ, Lin P, Tombal B, Saad F, Higano CS, Joshua AM, Parli T, Rosbrook B, van Os S, Beer TM. Five-year Survival Prediction and Safety Outcomes with Enzalutamide in Men with Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer from the PREVAIL Trial. Eur Urol. 2020 Sep;78(3):347-357. doi: 10.1016/j.eururo.2020.04.061. Epub 2020 Jun 9. PMID 32527692
- [Derived] Armstrong AJ, Al-Adhami M, Lin P, Parli T, Sugg J, Steinberg J, Tombal B, Sternberg CN, de Bono J, Scher HI, Beer TM. Association Between New Unconfirmed Bone Lesions and Outcomes in Men With Metastatic Castration-Resistant Prostate Cancer Treated With Enzalutamide: Secondary Analysis of the PREVAIL and AFFIRM Randomized Clinical Trials. JAMA Oncol. 2020 Feb 1;6(2):217-225. doi: 10.1001/jamaoncol.2019.4636. PMID 31830211
- [Derived] Armstrong AJ, Lin P, Higano CS, Iversen P, Sternberg CN, Tombal B, Phung D, Parli T, Krivoshik A, Beer TM. Prognostic Association of Prostate-specific Antigen Decline with Clinical Outcomes in Men with Metastatic Castration-resistant Prostate Cancer Treated with Enzalutamide in a Randomized Clinical Trial. Eur Urol Oncol. 2019 Nov;2(6):677-684. doi: 10.1016/j.euo.2018.11.005. Epub 2018 Dec 3. PMID 31274110
- [Derived] Armstrong AJ, Lin P, Higano CS, Sternberg CN, Sonpavde G, Tombal B, Templeton AJ, Fizazi K, Phung D, Wong EK, Krivoshik A, Beer TM. Development and validation of a prognostic model for overall survival in chemotherapy-naive men with metastatic castration-resistant prostate cancer. Ann Oncol. 2018 Nov 1;29(11):2200-2207. doi: 10.1093/annonc/mdy406. PMID 30202945
- [Derived] Rathkopf DE, Beer TM, Loriot Y, Higano CS, Armstrong AJ, Sternberg CN, de Bono JS, Tombal B, Parli T, Bhattacharya S, Phung D, Krivoshik A, Scher HI, Morris MJ. Radiographic Progression-Free Survival as a Clinically Meaningful End Point in Metastatic Castration-Resistant Prostate Cancer: The PREVAIL Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):694-701. doi: 10.1001/jamaoncol.2017.5808. PMID 29522174
- [Derived] Kim CS, Choi YD, Lee SE, Lee HM, Ueda T, Yonese J, Fukagai T, Chiong E, Lau W, Abhyankar S, Theeuwes A, Tombal B, Beer TM, Kimura G. Post hoc analyses of East Asian patients from the randomized placebo-controlled PREVAIL trial of enzalutamide in patients with chemotherapy-naive, metastatic castration-resistant prostate cancer. Medicine (Baltimore). 2017 Jul;96(27):e7223. doi: 10.1097/MD.0000000000007223. PMID 28682871
- [Derived] Devlin N, Herdman M, Pavesi M, Phung D, Naidoo S, Beer TM, Tombal B, Loriot Y, Ivanescu C, Parli T, Balk M, Holmstrom S. Health-related quality of life effects of enzalutamide in patients with metastatic castration-resistant prostate cancer: an in-depth post hoc analysis of EQ-5D data from the PREVAIL trial. Health Qual Life Outcomes. 2017 Jun 23;15(1):130. doi: 10.1186/s12955-017-0704-y. PMID 28645287
- [Derived] Bryce AH, Alumkal JJ, Armstrong A, Higano CS, Iversen P, Sternberg CN, Rathkopf D, Loriot Y, de Bono J, Tombal B, Abhyankar S, Lin P, Krivoshik A, Phung D, Beer TM. Radiographic progression with nonrising PSA in metastatic castration-resistant prostate cancer: post hoc analysis of PREVAIL. Prostate Cancer Prostatic Dis. 2017 Jun;20(2):221-227. doi: 10.1038/pcan.2016.71. Epub 2017 Jan 24. PMID 28117385
- [Derived] Beer TM, Armstrong AJ, Rathkopf D, Loriot Y, Sternberg CN, Higano CS, Iversen P, Evans CP, Kim CS, Kimura G, Miller K, Saad F, Bjartell AS, Borre M, Mulders P, Tammela TL, Parli T, Sari S, van Os S, Theeuwes A, Tombal B. Enzalutamide in Men with Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer: Extended Analysis of the Phase 3 PREVAIL Study. Eur Urol. 2017 Feb;71(2):151-154. doi: 10.1016/j.eururo.2016.07.032. Epub 2016 Jul 28. PMID 27477525
- [Derived] Kim CS, Theeuwes A, Kwon DD, Choi YD, Chung BH, Lee HM, Lee KH, Lee SE. The PREVAIL trial of enzalutamide in men with chemotherapy-naive, metastatic castration-resistant prostate cancer: Post hoc analysis of Korean patients. Investig Clin Urol. 2016 May;57(3):174-83. doi: 10.4111/icu.2016.57.3.174. Epub 2016 May 10. PMID 27195316
- [Derived] Graff JN, Baciarello G, Armstrong AJ, Higano CS, Iversen P, Flaig TW, Forer D, Parli T, Phung D, Tombal B, Beer TM, Sternberg CN. Efficacy and safety of enzalutamide in patients 75 years or older with chemotherapy-naive metastatic castration-resistant prostate cancer: results from PREVAIL. Ann Oncol. 2016 Feb;27(2):286-94. doi: 10.1093/annonc/mdv542. Epub 2015 Nov 16. PMID 26578735
- [Derived] Loriot Y, Miller K, Sternberg CN, Fizazi K, De Bono JS, Chowdhury S, Higano CS, Noonberg S, Holmstrom S, Mansbach H, Perabo FG, Phung D, Ivanescu C, Skaltsa K, Beer TM, Tombal B. Effect of enzalutamide on health-related quality of life, pain, and skeletal-related events in asymptomatic and minimally symptomatic, chemotherapy-naive patients with metastatic castration-resistant prostate cancer (PREVAIL): results from a randomised, phase 3 trial. Lancet Oncol. 2015 May;16(5):509-21. doi: 10.1016/S1470-2045(15)70113-0. Epub 2015 Apr 14. PMID 25888263
- [Derived] Beer TM, Armstrong AJ, Rathkopf DE, Loriot Y, Sternberg CN, Higano CS, Iversen P, Bhattacharya S, Carles J, Chowdhury S, Davis ID, de Bono JS, Evans CP, Fizazi K, Joshua AM, Kim CS, Kimura G, Mainwaring P, Mansbach H, Miller K, Noonberg SB, Perabo F, Phung D, Saad F, Scher HI, Taplin ME, Venner PM, Tombal B; PREVAIL Investigators. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014 Jul 31;371(5):424-33. doi: 10.1056/NEJMoa1405095. Epub 2014 Jun 1. PMID 24881730

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following the independent data monitoring committee's recommendation, a protocol amendment was implemented for double-blind phase to be proceeded to open-label phase, which allowed previously placebo treated participants who had not received commercial enzalutamide the opportunity, to receive open-label access to enzalutamide.
Groups:
- Enzalutamide: Participants received enzalutamide 160 mg, administered as four 40-mg capsules, once per day by mouth.
- Placebo: Participants received placebo, administered as four capsules, once per day by mouth.
- Placebo Participants Crossover to Enzalutamide: Participants who received placebo in double-blind period and who agreed to proceed to open-label phase period, received enzalutamide 160 mg, administered as four 40-mg capsules, once per day by mouth.
Period: Double-blind
Arm/Group | Enzalutamide | Placebo | Placebo Participants Crossover to Enzalutamide
Started | 872 | 845 | 0
Safety Population | 871 | 844 | 0
Completed | 0 | 234 | 0
Not Completed | 872 | 611 | 0
Not completed — Lost to Follow-up | 8 | 4 | 0
Not completed — Death | 699 | 550 | 0
Not completed — Withdrawal by Subject | 16 | 19 | 0
Not completed — Other | 7 | 0 | 0
Not completed — Sponsor decision | 142 | 38 | 0
Period: Open-label
Arm/Group | Enzalutamide | Placebo | Placebo Participants Crossover to Enzalutamide
Started | 0 | 0 (participants were given the opportunity to receive open-label access to enzalutamide) | 234 (previous placebo treated participants were given the opportunity to receive enzalutamide)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 234
Not completed — Death | 0 | 0 | 166
Not completed — Lost to Follow-up | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 7
Not completed — Sponsor decision | 0 | 0 | 53
Not completed — Other | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enzalutamide | Placebo | Total
Number analyzed (Participants) | 872 | 845 | 1717
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 179 | 179 | 358
  >=65 years | 693 | 666 | 1359
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (8.51) | 71.2 (8.42) | 71.3 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 872 | 845 | 1717
Region of Enrollment [Number; unit: count of participants]
  United States | 127 | 120 | 247
  Slovakia | 13 | 14 | 27
  Finland | 18 | 15 | 33
  Spain | 44 | 37 | 81
  Lithuania | 8 | 6 | 14
  Austria | 9 | 9 | 18
  Russian Federation | 12 | 10 | 22
  Israel | 14 | 11 | 25
  United Kingdom | 78 | 75 | 153
  Italy | 15 | 15 | 30
  France | 85 | 90 | 175
  Canada | 91 | 88 | 179
  Poland | 21 | 18 | 39
  Belgium | 28 | 29 | 57
  Singapore | 5 | 4 | 9
  Australia | 116 | 116 | 232
  Denmark | 43 | 44 | 87
  Netherlands | 15 | 13 | 28
  Germany | 41 | 42 | 83
  Japan | 28 | 33 | 61
  Sweden | 21 | 18 | 39
  Korea, Republic of | 40 | 38 | 78

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to death due to any cause. For patients who were alive at the time of the analysis data cutoff, overall survival was censored at the last date the patient was known to be alive or analysis data cutoff date, whichever was first. This included patients who were known to have died after the data analysis cutoff date. Patients with no post-baseline survival information were censored on the date of randomization.
Time Frame: During study period (up to 3 years)
Population: Intent to Treat (ITT) - All patients randomly assigned to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 872 | 845
months | 32.4 [30.1 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 30.2 [28.0 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — A 2-stage group sequential method (Lan DeMets OBF) assigned the level of significance for the pre-specified interim overall survival analysis (p<0.015) based on overall 2-sided type I error rate of 0.049. Final results based upon interim analysis; Hazard Ratio (HR) = 0.706, 95% CI 2-sided [0.596 to 0.837] — The hazard ratio is based on an unstratified Cox regression model (with treatment as the only covariate) and is relative to placebo with <1 favoring enzalutamide

2. Primary Outcome: Radiographic Progression-free Survival (rPFS)
Description: Radiographic progression-free survival was defined as the time from randomization to the first objective evidence of radiographic disease progression assessed by independent central radiology review or death due to any cause within 168 days after treatment discontinuation, whichever was first. Radiographic disease progression was evaluated by CT scan or MRI and radionuclide bone scans at regularly scheduled visits. Radiographic disease progression in bone required a confirmatory scan. Radiographic disease progression in soft tissue did not require a confirmatory scan for purposes of analysis. Radiographic disease progression was evaluated by independent central radiology review using RECIST 1.1 for soft tissue disease and PCWG2 guidelines for bone disease. Patients who did not reach the endpoint were censored at their last assessment.
Time Frame: During study period (up to 20 months)
Population: Intent to Treat (ITT) - All patients randomly assigned to treatment excluding 84 patients who were not randomized before the radiographic Progression-free Survival data cutoff date of 06 May 2012.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 832 | 801
months | NA [13.8 to NA] — The median time to radiographic progression-free survival and its upper 95% confidence limit were not yet reached in the enzalutamide group because an insufficient number of patients had an event at the time of analysis. | 3.9 [3.7 to 5.4]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — The assigned 2-sided type I error rate was 0.001 for the analysis of radiographic progression-free survival; Hazard Ratio (HR) = 0.186, 95% CI 2-sided [0.149 to 0.231] — The hazard ratio is based on an unstratified Cox regression model (with treatment as the only covariate) and is relative to placebo with < 1 favoring enzalutamide

3. Secondary Outcome: Time to First Skeletal-related Event
Description: Time to first skeletal-related event was defined as the time from randomization to the date of the first occurrence of a skeletal-related event for each patient. A skeletal-related event was defined as radiation therapy or surgery to bone for prostate cancer, pathological bone fracture, spinal cord compression, or initiation/change in antineoplastic therapy to treat bone pain from prostate cancer. Skeletal-related events were recorded at each scheduled and unscheduled study visit and during long-term follow-up if a skeletal-related event was not documented previously. Patients who did not have a skeletal-related event at the time of the analysis data cutoff were censored at the date of last assessment indicating no evidence of skeletal-related event. Patients with no postbaseline assessments were censored on the date of randomization.
Time Frame: During study period (up to 3 years)
Population: Intent to Treat (ITT) - All patients randomly assigned to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 872 | 845
months | 31.1 [29.5 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 31.3 [23.9 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — The Holm step down method of multiple comparisons was used to maintain a study wide type I error of 5% for prespecified secondary efficacy analyses. The 2-sided type I error rate was 0.01 for this analysis; Hazard Ratio (HR) = 0.718, 95% CI [0.610 to 0.844] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy
Description: The time to initiation of cytotoxic chemotherapy is defined as the time from randomization to the date of initiation of cytotoxic chemotherapy for the treatment of prostate cancer for each patient. For patients who did not start cytotoxic chemotherapy at the time of the analysis data cutoff, time to initiation of cytotoxic chemotherapy was censored at the date of last assessment where no cytotoxic chemotherapy was indicated or at the analysis data cutoff date, whichever was first. Time to initiation of cytotoxic chemotherapy for patients with no postbaseline assessments was censored on the date of randomization.
Time Frame: During study period (up to 3 years)
Population: Intent to Treat (ITT) - All patients randomly assigned to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 872 | 845
months | 28.0 [25.8 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 10.8 [9.7 to 12.2]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — The Holm step down method of multiple comparisons was used to maintain a study wide type I error of 5% for prespecified secondary efficacy analyses. The 2-sided type I error rate was 0.0125 for this analysis; Hazard Ratio (HR) = 0.349, 95% CI [0.303 to 0.403] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time to PSA progression was defined as the time from randomization to date of first confirmed observation of PSA progression for each patient. For patients with PSA declines at week 13, the PSA progression date was defined as the date that a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir was documented, and confirmed 3 or more weeks later. For patients with no PSA decline at week 13, the PSA progression date was defined as the date that a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above baseline was documented, and confirmed 3 or more weeks later. For patients who did not have confirmed PSA progression at the time of the analysis data cutoff, time to PSA progression was censored at the date of the last PSA assessment showing no evidence of confirmed PSA progression or the analysis data cutoff date, whichever was first. Time to PSA progression for patients with no postbaseline assessments was censored on the date of randomization.
Time Frame: During study period (up to 3 years)
Population: Intent to Treat (ITT) - All patients randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 872 | 845
months | 11.2 [11.1 to 13.7] | 2.8 [2.8 to 2.9]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — The Holm step down method of multiple comparisons was used to maintain a study wide type I error of 5% for prespecified secondary efficacy analyses. The 2-sided type I error rate was 0.0167 for this analysis; Hazard Ratio (HR) = 0.169, 95% CI [0.147 to 0.195] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percentage of Patients With Prostate Specific Antigen (PSA) Response ≥ 50%
Description: PSA response was defined as a ≥ 50% reduction in PSA from baseline to the lowest postbaseline PSA value and required confirmation by a consecutive assessment at least 3 weeks later. Patients were evaluable for PSA response rate if a patient had a PSA level measured at baseline and at least one postbaseline assessment.
Time Frame: During study period (up to 3 years)
Population: Evaluable intent to treat (ITT) population - All patients randomly assigned to treatment with PSA values at baseline and at least one postbaseline assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 854 | 777
Percentage of Participants | 78 [75.1 to 80.7] | 3.5 [2.3 to 5.0]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The Holm step down method of multiple comparisons was used to maintain a study wide type I error of 5% for prespecified secondary efficacy analyses. The 2-sided type I error rate was 0.025 for this analysis; Difference in response rates = 74.51, 95% CI [71.45 to 77.57]

7. Secondary Outcome: Best Overall Soft Tissue Response
Description: The best overall soft tissue objective response is defined as partial response [PR] or complete response [CR] while on study treatment based on investigator assessments of target, nontarget, and new lesions using RECIST 1.1. Soft tissue was assessed by CT or MRI at regularly scheduled visits. Only patients with measurable soft tissue disease (ie, at least 1 target lesion identified per RECIST 1.1) at screening are included in this analysis. All percentages are based on number of participants with measurable soft tissue disease at screening in each treatment group.
Time Frame: During study period (up to 3 years)
Population: Intent to treat (ITT) population With Measurable Disease - All participants who were randomly assigned to treatment and had at least one target lesion at screening.
Measure: Number; unit: Percentage of participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 396 | 381
Percentage of participants | 58.8 | 5.0
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The Holm step down method of multiple comparisons was used to maintain a study wide type I error of 5% for prespecified secondary efficacy analyses. The 2-sided type I error rate was 0.05 for this analysis; Difference in objective response rate = 53.85, 95% CI [48.53 to 59.17]

8. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to a maximum of 6.5 years that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline to discontinuation from the study or death, whichever occurred first (maximum duration of 6.5 years)
Population: The safety analysis set included all randomized participants who received at least 1 dose or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide | Placebo | Placebo Participants Crossover to Enzalutamide
Number analyzed (Participants) | 871 | 844 | 234
Participants
  AEs | 857 | 791 | 212
  SAEs | 384 | 229 | 104

9. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) Greater Than or Equal to (>=) Grade 3, Based on National Cancer Institute Common Terminology Criteria for AEs (CTCAE), Version 4.0
Description: An AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. As per NCI CTCAE, Grade 3 events =medically significant but not immediately life-threatening, unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment, Grade 4 events =participant to be in imminent danger of death. Grade 5 events =death. A treatment-emergent AE (TEAE) was defined as an AE that occurred from the date and time of the first dose of study drug up to a maximum duration of 6.5 years. Number of participants with AEs of any of the Grade 3 or above (Grade 4, 5) were reported.
Time Frame: Baseline to discontinuation from the study or death, whichever occurred first (maximum duration of 6.5 years)
Population: The safety analysis set included all randomized participants who received at least 1 dose or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide | Placebo | Placebo Participants Crossover to Enzalutamide
Number analyzed (Participants) | 871 | 844 | 234
Participants | 465 | 318 | 129

10. Other Pre Specified Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to a maximum duration of 6.5 years that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator.
Time Frame: Baseline to discontinuation from the study or death, whichever occurred first (maximum duration of 6.5 years)
Population: The safety analysis set included all randomized participants who received at least 1 dose or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide | Placebo | Placebo Participants Crossover to Enzalutamide
Number analyzed (Participants) | 871 | 844 | 234
Participants
  AEs | 579 | 423 | 119
  SAEs | 38 | 22 | 14

ADVERSE EVENTS:
Time Frame: Baseline to discontinuation from the study or death, whichever occurred first (maximum duration of 6.5 years)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis was performed on safety set.
Arm/Group | Enzalutamide | Placebo | Placebo Participants Crossover to Enzalutamide
All-Cause Mortality (participants affected / at risk) | 699/871 | 550/844 | 166/234
Serious Adverse Events (participants affected / at risk) | 384/871 | 229/844 | 104/234
Other Adverse Events (participants affected / at risk) | 814/871 | 723/844 | 180/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=871) | Placebo (N=844) | Placebo Participants Crossover to Enzalutamide (N=234)
Anaemia (Blood and lymphatic system disorders) | 18 | 9 | 6
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 10 | 6 | 0
Acute myocardial infarction (Cardiac disorders) | 11 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1 | 1
Atrioventricular block (Cardiac disorders) | 1 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 5 | 0 | 0
Angina pectoris (Cardiac disorders) | 3 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0
Amaurosis (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 15 | 10 | 6
Disease progression (General disorders) | 10 | 7 | 11
Death (General disorders) | 5 | 1 | 0
Oedema peripheral (General disorders) | 2 | 3 | 0
Fatigue (General disorders) | 5 | 0 | 2
Gait disturbance (General disorders) | 2 | 1 | 0
Pain (General disorders) | 3 | 0 | 0
Performance status decreased (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 1 | 3
Asthenia (General disorders) | 0 | 1 | 5
Chest pain (General disorders) | 1 | 0 | 0
Device dislocation (General disorders) | 1 | 1 | 1
Drowning (General disorders) | 1 | 0 | 0
Generalized oedema (General disorders) | 1 | 0 | 0
Medical device complication (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0
Suprapubic pain (General disorders) | 0 | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0
Device occlusion (General disorders) | 2 | 1 | 0
Local swelling (General disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 14 | 7 | 8
Urinary tract infection (Infections and infestations) | 8 | 5 | 10
Urosepsis (Infections and infestations) | 5 | 3 | 4
Sepsis (Infections and infestations) | 3 | 4 | 1
Gastroenteritis (Infections and infestations) | 4 | 1 | 0
Device related infection (Infections and infestations) | 2 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0
Gallbladder abscess (Infections and infestations) | 0 | 1 | 0
Gastroenteritis staphylococcal (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 12 | 3 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 7 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 4 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 2 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 2 | 0
Arteriogram coronary (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Coagulation time prolonged (Investigations) | 1 | 0 | 0
Eastern cooperative oncology group performance status worsened (Investigations) | 0 | 1 | 0
International normalized ratio increased (Investigations) | 0 | 1 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 15 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 | 2 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 17 | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer limited stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 35 | 25 | 10
Syncope (Nervous system disorders) | 8 | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 7 | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 4 | 0 | 0
Nerve root compression (Nervous system disorders) | 2 | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 6 | 3 | 0
Presyncope (Nervous system disorders) | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0
Paraparesis (Nervous system disorders) | 1 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Coma hepatic (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Meningorrhagia (Nervous system disorders) | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 1 | 0
Spinal cord ischaemia (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0 | 0
Vith nerve disorder (Nervous system disorders) | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 4 | 2
Suicide attempt (Psychiatric disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 10 | 13 | 3
Haematuria (Renal and urinary disorders) | 11 | 12 | 3
Urinary tract obstruction (Renal and urinary disorders) | 8 | 9 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 11 | 1
Renal failure acute (Renal and urinary disorders) | 6 | 5 | 2
Ureteric obstruction (Renal and urinary disorders) | 4 | 4 | 1
Obstructive uropathy (Renal and urinary disorders) | 5 | 6 | 3
Bladder outlet obstruction (Renal and urinary disorders) | 2 | 3 | 0
Postrenal failure (Renal and urinary disorders) | 2 | 3 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 3 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 1 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tracheal obstruction extrinsic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cancer hormonal therapy (Surgical and medical procedures) | 1 | 0 | 0
Pain management (Surgical and medical procedures) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 2 | 0
Hypertension (Vascular disorders) | 4 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 2 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 0
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Platelet Dysfunction (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 0 | 2
Atrial Tachycardia (Cardiac disorders) | 0 | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 3 | 2 | 0
Cardiac Failure (Cardiac disorders) | 5 | 2 | 3
Cardiac Failure Congestive (Cardiac disorders) | 2 | 1 | 1
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0 | 0
Cardiovascular Insufficiency (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 6 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 0 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 2 | 0 | 0
Mitral Valve Disease (Cardiac disorders) | 1 | 0 | 0
Mitral Valve Incompetence (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 6 | 1 | 1
Supraventricular Tachycardia (Cardiac disorders) | 2 | 0 | 1
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 1 | 0 | 0
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 1 | 0 | 0
Eyelid Ptosis (Eye disorders) | 1 | 0 | 0
Retinal Vein Occlusion (Eye disorders) | 1 | 0 | 0
Anal Stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal Spasm (Gastrointestinal disorders) | 1 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Device Malfunction (General disorders) | 1 | 0 | 0
Medical Device Pain (General disorders) | 0 | 1 | 0
Multi-Organ Failure (General disorders) | 3 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic Cyst (Hepatobiliary disorders) | 1 | 0 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0 | 0
Cholecystitis Infective (Infections and infestations) | 1 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 1
Clostridium Difficile Sepsis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Infected Dermal Cyst (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 2 | 0 | 3
Meningitis Pneumococcal (Infections and infestations) | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0 | 0
Pulmonary Sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2
Back Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Bile Leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Renal Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sternal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Biopsy (Investigations) | 1 | 0 | 0
Ejection Fraction Decreased (Investigations) | 1 | 0 | 0
Electrocardiogram Abnormal (Investigations) | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases To Chest Wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases To Penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cervical Cord Compression (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 1
Cranial Nerve Paralysis (Nervous system disorders) | 1 | 0 | 0
Grand Mal Convulsion (Nervous system disorders) | 1 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0 | 1
Neurological Symptom (Nervous system disorders) | 1 | 0 | 0
Sensory Loss (Nervous system disorders) | 0 | 0 | 1
Vith Nerve Paralysis (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Epiduritis (Nervous system disorders) | 0 | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Knee Arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Radical Cystectomy (Surgical and medical procedures) | 0 | 0 | 1
Umbilical Hernia Repair (Surgical and medical procedures) | 1 | 0 | 0
Aneurysm (Vascular disorders) | 1 | 0 | 0
Peripheral Artery Stenosis (Vascular disorders) | 1 | 0 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 2 | 0 | 0
Status Epilepticus (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=871) | Placebo (N=844) | Placebo Participants Crossover to Enzalutamide (N=234)
Anaemia (Blood and lymphatic system disorders) | 76 | 68 | 23
Nausea (Gastrointestinal disorders) | 211 | 192 | 34
Constipation (Gastrointestinal disorders) | 220 | 145 | 38
Diarrhoea (Gastrointestinal disorders) | 160 | 121 | 20
Vomiting (Gastrointestinal disorders) | 64 | 70 | 9
Abdominal pain (Gastrointestinal disorders) | 56 | 31 | 4
Fatigue (General disorders) | 332 | 220 | 63
Asthenia (General disorders) | 122 | 69 | 15
Oedema peripheral (General disorders) | 115 | 70 | 20
Urinary tract infection (Infections and infestations) | 70 | 56 | 11
Nasopharyngitis (Infections and infestations) | 74 | 44 | 6
Upper respiratory tract infection (Infections and infestations) | 61 | 30 | 7
Fall (Injury, poisoning and procedural complications) | 136 | 42 | 15
Weight decreased (Investigations) | 122 | 72 | 26
Decreased appetite (Metabolism and nutrition disorders) | 182 | 139 | 36
Back pain (Musculoskeletal and connective tissue disorders) | 280 | 188 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 206 | 137 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 124 | 97 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 100 | 116 | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 112 | 74 | 28
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 73 | 40 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 59 | 49 | 8
Headache (Nervous system disorders) | 102 | 59 | 15
Dizziness (Nervous system disorders) | 85 | 54 | 13
Dysgeusia (Nervous system disorders) | 67 | 31 | 5
Insomnia (Psychiatric disorders) | 78 | 48 | 10
Haematuria (Renal and urinary disorders) | 93 | 43 | 11
Pollakiuria (Renal and urinary disorders) | 62 | 37 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 95 | 58 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 88 | 60 | 14
Hot flush (Vascular disorders) | 159 | 66 | 11
Hypertension (Vascular disorders) | 148 | 36 | 28
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 45 | 27 | 8
Rash (Skin and subcutaneous tissue disorders) | 31 | 21 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees not to independently publish the results before the publication of the multi-center PI paper. Sponsor shall review and comment 30 days prior to submission or disclosure. If publication or disclosure contains Sponsor Confidential Information, other than study data, PI agrees to remove Confidential Information from publication or disclosure. Sponsor may request that PI delay such publication for an additional 60 days to protect the patentability of any invention described.